CLINICAL TRIAL: NCT00310466
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Parallel Group Clinical Trial to Investigate the Efficacy and Safety of Specific Sublingual Immunotherapy With SLITone Birch in Patients With Seasonal Birch Pollen Induced Rhinoconjunctivitis
Brief Title: Efficacy and Safety Trial of SLITone(TM) Birch in Subjects With Hayfever
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHX0712
Record Dates: First submitted 2006-04-02; First posted 2006-04-04 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-04

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual immunotherapy (Active Comparator): sublingual immunotherapy with drops applied once daily by single dose containers (200 STU per dose)
  Interventions: Biological: Sublingual immunotherapy
- Placebo (Placebo Comparator): placebo sublingual drops
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Sublingual immunotherapy — once daily intake of sublingual drops
  Other Names: SLITone(TM) Birch
  Arms: Sublingual immunotherapy
Biological: Placebo — once daily intake of sublingual drops
  Arms: Placebo

SUMMARY:
The trial is performed to assess the efficacy and safety of SLIT One birch for treatment of birch pollen induced allergy

DETAILED DESCRIPTION:
Daily rhinoconjunctivits symptom and medication scores from patient diaries, adverse events

ELIGIBILITY:
Inclusion Criteria:

* A history of birch pollen allergy
* Positive skin prick test to birch
* Positive conjunctival test to birch
* Positive specific Immunoglobulin E (IgE) to birch

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1)<70% of predicted value
* History of seasonal allergy interfering with study
* History of symptomatic perennial allergy
* History of emergency visit or admission for asthma in the previous 12 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Wolf, PhD, Study Director — ALK-SCHERAX Arzneimittel GmbH; Margitta Worm, MD, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Klinik für Dermatologie, Venerologie und Allergologie, Berlin, State of Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 13 June 2005
Groups:
- SLITone Birch: Birch pollen extract for sublingual administration
- Placebo: Corresponding placebo for sublingual administration
Period: Overall Study
Arm/Group | SLITone Birch | Placebo
Started | 113 | 113
Completed | 95 | 101
Not Completed | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLITone Birch | Placebo | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 113 | 113 | 226.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.9) | 39.5 (11.5) | 39.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 71 | 140.0
  Male | 44 | 42 | 86.0
Region of Enrollment [Number; unit: participants]
  Germany | 113 | 113 | 226.0

OUTCOME MEASURES:

1. Primary Outcome: Daily Rhinoconjunctivitis Symptom Score
Description: A total of 6 rhinoconjunctivitis symptoms are recorded (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes, watery eyes). Each symptoms is scored on a scale from 0-3 (no symptoms-severe symptoms). I.e. the total daily score can be 0-18.
Time Frame: Birch pollen season 2006
Measure: Mean (Standard Deviation); unit: Units on a scale (0-18)
Arm/Group | SLITone Birch | Placebo
Number analyzed (Participants) | 95 | 101
Units on a scale (0-18) | 4.07 (2.59) | 4.14 (2.56)
Statistical Analysis 1: Comparison: SLITone Birch vs Placebo; Test type: Superiority or Other; p = 0.87, ANOVA

2. Secondary Outcome: Global Improvement of Rhinoconjunctivitis Symptoms Assessed by the Subjects
Description: The number of participants who reported improved overall symptoms compared to the previous birch pollen season (each patient was asked to compare his/her symptoms in the 2006 birch pollen season with the symptoms in the 2005 birch pollen season).
Time Frame: Birch pollen season 2006
Measure: Number; unit: Participants
Arm/Group | SLITone Birch | Placebo
Number analyzed (Participants) | 95 | 101
Participants | 48 | 42
Statistical Analysis 1: Comparison: SLITone Birch vs Placebo; Test type: Superiority or Other; p = 0.04, ANOVA

3. Secondary Outcome: Adverse Events
Description: An adverse event was defined as: Any untoward medical occurence in a patient or clinical trial subject administered a trial product and which does not necessarily have a causal relationship with this treatment (International Conference of Harmonisation (ICH) Harmonised Tripartite Guideline E2A, Step 5).
Time Frame: Birch pollen season 2006
Measure: Number; unit: Events
Arm/Group | SLITone Birch | Placebo
Number analyzed (Participants) | 95 | 101
Events | 81 | 87

4. Primary Outcome: Daily Rhinoconjunctivitis Rescue Medication Score
Description: Rescue medication (desloratadine tablets, budesonide nasal spray, prednisone tablets) used for treatment of rhinoconjunctivitis symptoms not controlled by the study medication, were recorded. The total daily score was 0-30 (No medication-Maximum use of medication).
Time Frame: Birch pollen season 2006
Measure: Mean (Standard Deviation); unit: Units on a scale (0-30)
Arm/Group | SLITone Birch | Placebo
Number analyzed (Participants) | 95 | 101
Units on a scale (0-30) | 2.76 (3.30) | 2.54 (2.99)
Statistical Analysis 1: Comparison: SLITone Birch vs Placebo; Test type: Superiority or Other; p = 0.55, ANOVA

ADVERSE EVENTS:
Arm/Group | SLITone Birch | Placebo
Serious Adverse Events (participants affected / at risk) | 4/113 | 2/113
Other Adverse Events (participants affected / at risk) | 81/113 | 87/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLITone Birch (N=113) | Placebo (N=113)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLITone Birch (N=113) | Placebo (N=113)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Arrhytmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (5) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 8 (10) | 7 (8)
Eye redness (Eye disorders) | 0 (0) | 3 (3)
Eye swelling (Eye disorders) | 2 (3) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 11 (14) | 7 (8)
Oral pruritus (Gastrointestinal disorders) | 37 (45) | 27 (31)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Application site anaesthesia (General disorders) | 0 (0) | 1 (1)
Application site eczema (General disorders) | 0 (0) | 1 (1)
Application site papules (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 2 (2)
Mucous membrane disorders (General disorders) | 0 (0) | 1 (1)
Oedema mucosal (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sensation of foreign body (General disorders) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (4)
Seasonal allergy (Immune system disorders) | 2 (3) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 4 (6)
Cystitis (Infections and infestations) | 1 (1) | 2 (3)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes soster (Infections and infestations) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2)
Infected naevus (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (6)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis viral (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (17) | 15 (16)
Otitis media (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 3 (4)
Rhinitis infective (Infections and infestations) | 0 (0) | 2 (2)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (5) | 5 (5)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Vaginitis (Infections and infestations) | 0 (0) | 1 (1)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Bone spur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Oral dysaesthesia (Nervous system disorders) | 3 (3) | 3 (3)
Paraesthesia oral (Nervous system disorders) | 13 (17) | 6 (8)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (6)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Maxillary sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (4)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis medicamentosa (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Exanthem (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Dental operation (Surgical and medical procedures) | 1 (2) | 1 (1)
Joint surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Clinical improvement following SLIT is thought to be due to immunological mechanisms that develop over time. Even though clear immunological changes were observed in this trial it appears that the treatment was too short to reach full clinical effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ALK must receive copies of any intended communication in advance of publication (at least 15 working days for an abstract or oral presentation and 45 working days for a journal submission). ALK will review the communications for accuracy (thus avoiding potential discrepancies with submissions to health authorities), verify that confidential information is not being inadvertently divulged and provide any relevant supplementary information.